CLINICAL TRIAL: NCT04850053
Title: Detection of Alzheimer's Disease (AD)-Related Seeds as Biomarkers for Accurate Diagnosis of AD（AD-seeds-detector）
Brief Title: Detection of Alzheimer's Disease (AD)-Related Seeds for AD Diagnosis
Status: Recruiting | Type: Observational
Sponsor: Capital Medical University (Other)
Collaborators: Shandong Provincial Hospital (Other Government); Xiangya Hospital of Central South University (Other); Zhejiang Provincial People's Hospital (Other); Beijing Geriatric Hospital (Other); Kaifeng Central Hospital (Other); The First Affiliated Hospital of Chongqing Medical Universty (Unknown); Huashan Hospital (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); West China Hospital (Other); Henan Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Jianping Jia, Chief Director, Capital Medical University
Other Study IDs: AD-seeds-detector
Record Dates: First submitted 2021-04-14; First posted 2021-04-20 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood,cerebral spinal fluid
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Alzheimer's disease: Criteria for AD according to the 2011 NIA-AA
- Non-AD dementia: Frontotemporal dementia (FTD); or Parkinson's disease dementia (PDD); or dementia with Lewy bodies (DLB); or vascular dementia (VaD); or corticobasal degeneration (CBD); or dementia not otherwise specified.
- Cognitively normal controls: Individuals with normal cognitive function

SUMMARY:
The study will investigate the biomarkers of Aβ and Tau seeds in plasma detected by Alzheimer's disease (AD) related seeds quantitative detector (AD-seeds-detector), and their sensitivity and specificity in diagnosing AD, compared with those from age-matched cognitively normal controls, and those with other types of dementia.

To perform a high throughput analysis of the amount of Aβ and Tau seeds, the investigators have developed an AD-seeds-detector, in which a fluorescence microplate reader was combined with an oscillating mixer or water-bath-type ultrasonicator.

DETAILED DESCRIPTION:
Aβ and Tau seeds have the potential to serve as biomarkers for AD. The AD-seeds-detector could detect small quantities of Aβ and Tau seeds by taking advantage of their ability to nucleate and enhance aggregation, enabling a very high amplification of the signal. This study examines the effectiveness of using the AD-seeds-detector as a novel technique for discriminating AD from cognitively normal control and non-AD dementia by detecting small Aβ and Tau seeds in plasma.

This will be an observational study aiming at using the AD-seeds-detector to detect minute amounts of Aβ and Tau seeds in plasma as novel biomarkers with high sensitivity and specificity for the accurate diagnosis of AD. To achieve this goal, the investigators will conduct two studies using the AD-seeds-detector to detect the Aβ and Tau seeds in the plasma samples.

Study one:

A single-center cohort that consists of well-characterized AD patients (n=150), cognitively normal controls (n=100) and non-AD dementia patients (n=50).

Study two:

A multi-center cohort with well-characterized AD patients (n=400), cognitively normal controls (n=400) and non-AD dementia patients (n=400).

ELIGIBILITY:
Inclusion Criteria:

* Aged 55-75. Written informed consent obtained from participant or legal guardian prior to any study-related procedures. The diagnosis of AD is made using the National Institute on Aging and the Alzheimer's Association (NIA-AA) criteria. As for non-AD dementia, the McKeith criteria are used for DLB,the revised diagnostic criteria proposed by the International behavioral variant (bvFTD) Criteria Consortium for bvFTD,the Gorno-Tempini criteria for the semantic variant FTD or non-fluent aphasia, the Movement Disorder Society Task Force criteria for PDD, the vascular behavioral and cognitive disorders (Vas-Cog) criteria for VaD, the Armstrong's criteria for CBD, the CDC's diagnostic criteria for CJD, etc. In addition, normal cognition is supported by MMSE, CDR and other cognitive function scales.

Exclusion Criteria:

* Other medical or psychiatric illness. No one can serve as an informant. Refused to complete a cognitive test and provide biospecimen.

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study one: (1) AD patients (n=150); (2) cognitively normal controls (n=100); (3) non-AD dementia patients (n=50).
  Study two: (1) AD patients (n=400); (2) cognitively normal controls (n=400); (3) non-AD dementia patients (n=400).
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2020-08-26 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The area under curve of the AD-seeds-detector for the accurate diagnosis of AD | two years
  The area under curve is used to show the ability of the AD-seeds-detector to diagnose AD. The value of area under curve is higher, then the ability of the AD-seeds-detector to diagnose AD is stronger.

SECONDARY OUTCOMES:
The sensitivity | two years
  The sensitivity is used to show the ability of the AD-seeds-detector to diagnose AD patients, and is represented by true positive/ (true positive +false negative).
The specificity | two years
  The specificity is used to show the ability of the AD-seeds-detector to avoid false AD patients and rule out AD patients, and is represented by true negative/ (false positive + true negative).
The positive predictive value | two years
  The positive predictive value is used to show the ability of the AD-seeds-detector to correctly label AD patients who test positive, and is represented by true positive / (true positive + false positive)
The negative predictive value | two years
  The negative predictive value is used to show the ability of the AD-seeds-detector to correctly label people who test negative, and is represented by true negative / (false negative + true negative)
Cellular toxcity of Aβ seeds protein | two years
  Toxcity of Aβ seeds protein on cells
Morphology and structure of Aβ | two years
  Comparison of Morphology and structure of beta-amyloid protein between difference groups

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital of Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jia J, Li T, Yang J, Chen B, Qin W, Wei C, Song Y, Wang Q, Li Y, Jia L. Detection of plasma Abeta seeding activity by a newly developed analyzer for diagnosis of Alzheimer's disease. Alzheimers Res Ther. 2022 Feb 2;14(1):21. doi: 10.1186/s13195-022-00964-2. PMID 35109911